CLINICAL TRIAL: NCT05187520
Title: Efficacy of Epidural Analgesia Versus Single Dose Injection of Naldebain® in Management of Acute and Chronic Surgical Pain After Cesarean Section in Term Parturient - a PI-initiated, Randomized, Open-label, Non-inferiority Clinical Trial
Brief Title: Naldebain for Control of Post-Cesarean Section Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: E-DA Hospital (Other)
Responsible Party: Principal Investigator, Tu, Yuan-Kun, Clinical Professor and Superintendent, E-DA Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMRP05111N
Record Dates: First submitted 2021-12-24; First posted 2022-01-11 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Post Operative Pain, Acute; Post Operative Pain, Chronic; Cesarean Section
Keywords: Epidural analgesia; Multimodal analgesia; Opioid use; Epidural analgesia complications; Quality of life
MeSH Terms: conditions — Pain, Postoperative | interventions — sebacoyl dinalbuphine ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-controlled epidural analgesia (PCEA) (Active Comparator): Patients assigned to PCEA group will receive epidural analgesia as the standard postoperative pain control strategy. After completion of cesarean section, a PCEA device will be connected to the epidural catheter to deliver mixture of local anesthetic (0.8 mg/ml) and fentanyl (2 mcg/ml) with preset continuous dose of 3-5 ml/h and a bolus dose of 3-4 ml.
  Interventions: Device: Patient-controlled epidural analgesia (PCEA)
- Naldebain® (Experimental): Patients assigned to Naldebain® group will receive a single intramuscular injection of dinalbuphine sebacate (150 mg in 2 ml solvent containing benzyl benzoate and sesame oil) into the gluteus muscles under ultrasound-guidance after completion of cesarean section.
  Interventions: Drug: Naldebain®

INTERVENTIONS:
Device: Patient-controlled epidural analgesia (PCEA) — Epidural analgesia is a technique of neuraxial block by placement of a 20G polyether epidural catheter into the epidural lumen and fixed at the desired depth, and analgesic effect is usually achieved by administration of mixture of local anesthetics and opioids using a programmed pump.
  Arms: Patient-controlled epidural analgesia (PCEA)
Drug: Naldebain® — Naldebain dissolved in benzyl benzoate and sesame oil (a total volume of 2ml) will be prepared in a 5-ml syringe 30 min before administration. Intramuscular injection into the gluteal muscles will be performed by an anesthesiologist under sonography-guidance.
  Other Names: Naldebain ER®; Sebacoyl Dinalbuphine Ester Injection
  Arms: Naldebain®

SUMMARY:
Inadequate postoperative pain management can lead to physical and psychological distress in patients as well as impact surgical wound healing and increase the risk of developing postoperative delirium and cardiopulmonary and thromboembolic events. Severe postoperative pain may also result in the development of chronic post-surgical pain (CPSP), which in turn can lead to prolonged use of opioids and increased health-care costs. A descriptive survey study in 60 postpartum women who received cesarean section suggested that the presence of postoperative pain significantly reduced the willingness of breastfeeding and infant care. The incidence of CPSP after cesarean delivery has been reported to vary from 1% to 18% up to 1 year after operation. Patient-controlled epidural analgesia (PCEA) is considered as the standard pain management strategy for post-cesarean pain. However, correct placement of epidural catheter for effective postoperative pain management is more technical demanding, and accidental dural puncture is associated with increased risk of postdural puncture headache. It also increases risk of other complications, including urinary retention, systemic toxicity of local anesthetics and formation of epidural hematoma. Therefore, the development of a safe, conveniently operated, and long-lasting analgesic strategy, which serves as background pain control modality up to several days after cesarean section should provide clinically beneficial advantages in the management of acute postoperative pain and prevention of CPSP in postpartum women. Naldebain® is prodrug of nalbuphine, which was approved by the Taiwan FDA in 2017. Naldebain® is rapidly hydrolyzed by tissue of plasma esterase to release nalbuphine. The bioavailability of nalbuphine following intramuscular injection Naldebain® was 85.4%, and it took approximately 6 days for the complete release of Naldebain® into the blood circulation. Therefore, a single parenteral injection of Naldebain® could provide long lasting analgesic effect in several phase II trials. However, Naldebain® has not been tested in the pain control after cesarean section. Therefore, this PI-initiated prospective, randomized, open-label, non-inferiority trial aims to investigate the clinical efficacy of Naldebain® in management of acute postoperative pain in term parturient who receive elective cesarean section to provide analgesic effect that is not inferior to the standard PCEA and prevent the development of CPSP.

DETAILED DESCRIPTION:
Inadequate postoperative pain management can lead to physical and psychological distress in patients as well as impact surgical wound healing and increase the risk of developing postoperative delirium and cardiopulmonary and thromboembolic events. Severe postoperative pain may also result in the development of chronic pain, which in turn can lead to prolonged use of opioids and increased health-care costs. Although clinical pathways and strategies have been recently implemented, including the introduction of the enhanced recovery after surgery (ERAS) program and multimodal analgesia (MMA), rates of inadequate postoperative pain management remain as high as 40-56.4% in the general surgical population and the prevalence rates of persistent pain after major operations can reach up to 50%. CPSP is associated with increased analgesic use, restriction of activities of daily living, significant effects on quality of life, and increased health-care utilization.

According to the WHO survey in 2004, cesarean section deliveries represent up to 8% of all surgical procedures. In Taiwan, about 35.9% of the newborns were delivered by cesarean section in 2016 to 2019, which equivalent to 68,000 cesarean sections were underwent annually. The incidence of CPSP after cesarean delivery has been reported to vary from 1% to 18% up to 1 year after operation. More specifically, an US nationwide survey reported that 79% of mothers who received cesarean section reported experiencing pain at the incision site in the first two months and 18% had persistent pain at least 6 months after operation. Following surgical incision of abdominal wall and visceral organs, the efferent sensory neurons initiate the cascade of neurochemical changes that activates and sensitizes the peripheral nociceptors and spinal dorsal horn neurons, leading to peripheral and central sensitization and a hyperalgesic state. With inadequate pain management after operation or prolonged healing process, the sustained activation of the pronociceptive system results in hyperalgesia and allodynia. Surgical insults and neuron axon damage may also activate regional inflammatory and immune reactions to release of neurotransmitters in the spinal cord to produce hypersensitivity and ectopic neural activity, and eventually contributing to the development of central sensitization and CPSP.

At the beginning 3-6 months, the incisional wound and abdomen are the most commonly reported location of persisted pain, and the unpleasant feeling shifts to the back or low back at 12 months postpartum and the chronic pain may significantly impact the quality of life, as one-fifth of patients complain of moderate to very severe pain. A prospective observational study found that the presence of CPSP after cesarean section negatively impacted the daily activity, normal work, social relationship, psychosomatic status and postpartum depression of the mothers at 3-6 months after delivery. A descriptive survey study in 60 postpartum women who received cesarean section suggested that the presence of postoperative pain significantly reduced the willingness of breastfeeding and infant care. Previous reports identified several important risk factors for developing CPSP after cesarean section, including previous cesarean delivery, preoperative depression or anxiety, lower society economic status, longer duration of surgery and use of general anesthesia. Most importantly, substantial evidence indicates that supports the general concept that higher severity of acute pain after cesarean section is associated with significantly higher risk for transition of acute pain to CPSP. Therefore, optimal but adequate pain management after cesarean section is important to improve postpartum care, accelerate recovery after surgery, enhance early mobilization and prevent the development of CPSP.

Multimodal analgesia (MMA) is the core principle for pain management after cesarean delivery, including epidural analgesia, the use of long-acting intrathecal opioids (i.e. morphine), and adjunct drugs (acetaminophen and nonsteroidal anti-inflammatory drugs). Intrathecal morphine is considered as the gold standard single-shot drug for post-cesarean pain, providing adequate analgesic effect up to 14-36h after operation. Placement of an epidural catheter can be used for epidural anesthesia during cesarean section and continuous epidural infusions of opioids or combined with local anesthetic after cesarean section can result in high-quality analgesia effect for postpartum and postsurgical pain. Compared with intrathecal morphine (ITM) alone, levels of pain scores both at rest and during mobilization were significantly reduced in women who received patient controlled epidural analgesia (PCEA) during the second day after cesarean section. Incidence of postoperative nausea and vomiting was also significantly lower in the PCEA group. A more recent randomized control trial reported that combination of PCEA with ITM provided better post-cesarean section analgesia compared to ITM alone. Although PCEA provides with patient-controlled, better analgesic effect, particularly the management of breakthrough pain or pain during mobilization, PCEA carries certain clinical concerns that impede their widely use in pain management after cesarean section. Correct placement of epidural catheter for effective postoperative pain management is more technical demanding, and accidental dural puncture is associated with increased risk of postdural puncture headache (PDPH). The most common complication of PCEA is urinary retention, especially when high concentrations of local anesthetic are used. The overall incidence of epidural hematoma and epidural abscess were 1 case per 168,000 and 1 per 145,000 women, respectively. Most seriously, unintentional intrathecal injection of large doses of local anesthetic can result in high spinal blocks, leading to respiratory compromise, and unintentional intravenous injection of local anesthetics can cause severe systemic toxicity, including seizures and cardiac arrest. Therefore, the development of a safe, conveniently operated, and long-lasting analgesic strategy, which serves as background pain control modality up to several days after cesarean section should provide clinically beneficial advantages in the management of acute postoperative pain and prevention of development of CPSP in postpartum women.

Nalbuphine is a synthetic agonist-antagonist opioid with analgesic properties acting on antagonism at the μ-receptor and agonism at the κ-receptor that was introduced for medical use in 1979. Nalbuphine has equal potency with morphine for pain relief, but it is associated with less nausea, pruritus, and respiratory depression than morphine due to its effect on κ-receptor. Since it is also a weak μ-receptor antagonist, nalbuphine reduces side effects particularly respiratory depression without loss of analgesia when combined with potent opioids. The other major clinical advantage of nalbuphine is less risk for abuse and death due to its ceiling effect of analgesia and respiratory suppression. Nalbuphine is one of the systemic administered opioids that can be safely used and effectively reduce the incisional pain and uterine cramping pain in women after cesarean section. Breast-feeding is also permissible when nalbuphine is administered to the mother to treat postpartum pain, as very low oral bioavailability of nalbuphine and the relative infant dose is 0.59+/-0.27% of the weight-adjusted maternal daily dose. However, the clinical use of nalbuphine for post-cesarean section pain control is limited by the relatively short duration of action of about 2-6h following systemic injection.

Naldebain® is prodrug of nalbuphine, which was approved by the Taiwan FDA in 2017. Naldebain® is an extended-release dinalbuphine sebacate, and is rapidly hydrolyzed by tissue of plasma esterase to release nalbuphine. The bioavailability of nalbuphine following intramuscular injection Naldebain® was 85.4% with a mean absorption time up to 145 h, and it took approximately 6 days for the complete release of Naldebain® into the blood circulation. Therefore, a single parenteral injection of Naldebain® could theoretically provide long lasting analgesic effect. The first clinical trial testing the perioperative analgesic effect of Naldebain® was reported in patients who received hemorrhoidectomy at 6 medical centers in Taiwan. 221 patients were randomly assigned to receive Naldebain® or vehicle injection at 1 day before operation. The average pain intensity scores (AUC of VAS) over 48h and 7 days after hemorrhoidectomy were significantly reduced in Naldebain® group (209.93 vs. 253.53 and 630.79 vs. 749.94, respectively). The Naldebain® group also had significantly lower doses of rescue analgesics. Furthermore, most adverse events were assessed as mild and tolerable in patients who received Naldebain® or the vehicle solution (benzyl benzoate and sesame oil). Most recently, a prospective, open-label, randomized controlled study was performed in 110 patients scheduled for elective laparotomy. The results showed that preoperative injection Naldebain® (150 mg) significantly reduce AUC of VAS at 4, 24, 32, 72, 120, and 144 h after surgery with a better quality of life during the recovery phase. A retrospective study analyzed the pain intensities in 137 patients who underwent midline laparotomy for gynecologic cancers and reported that a single intramuscular (IM) injection of Naldebain® significantly reduced the pain intensities than the fentanyl-based patient-controlled analgesia and conventional analgesia groups on postoperative days 1 to 5 with less analgesic-related side effects. The most commonly reported drug-related adverse reactions of Naldebain® are generally well tolerable, including dizziness (6-27%), nausea/vomiting (3-30%), injection site reactions (1.8-12%) and pyrexia.35-37 Hence, a single-dose IM administration of Naldebain® can be served as an effective long-acting preventive analgesic as a component of MMA that can enhance postoperative pain management and attenuate the development of CPSP.

Naldebain® has not been tested in the pain control after cesarean section and its pharmacokinetic profiles in the milk excretion of lactating women was also undetermined. Therefore, this PI-initiated prospective, randomized, open-label, non-inferiority trial aims to investigate the clinical efficacy of Naldebain® in management of acute postoperative pain in term parturient who receive elective cesarean section, and prevention of the development of CPSP after cesarean delivery, as Naldebain® can provide prolonged analgesic effect for up to 7 days. This study will also analyze the milk-plasma levels of nalbuphine following a single intramuscular injection in the parturient.

Null hypothesis: the investigators hypothesize that a single-dose IM injection of Naldebain® (alternative treatment) is inferior to PCEA (standard treatment) for controlling pain after cesarean section. The alternative hypothesis: a single-dose IM injection of Naldebain® (alternative treatment) is non-inferior to PCEA (standard treatment) for controlling pain after cesarean section. The study defines a non-inferiority margin of 10% difference in the average pain score (0-10) at postoperative days 1-3 in Naldebain® (alternative treatment) and PCEA (standard treatment) groups. The investigators speculated a P-value <0.05 indicates non-inferiority of a single-dose IM injection of Naldebain® to manage pain intensity after cesarean section in postpartum women in comparison to the standard PCEA, corresponding to the upper limit of the one-sided 95% confidence interval (CI) of the difference not exceeding the 10% based on the type I error at 0.05 (one-sided) and a 90% statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Term primipara or multipara

Exclusion Criteria:

* Severe pregnancy-induced complication (such as preeclampsia, eclampsia, poorly control pregnancy-induced hypertension and/or diabetes)
* High risk for postpartum hemorrhage
* Contraindications for neuraxial block
* Preterm (gestational age< 36 week) delivery
* Emergency cesarean section
* After-office hour schedule
* History of substance abuse
* Known allergy to nalbuphine, benzyl benzoate or sesame oil
* Not willing to follow the assignment of treatment after randomization

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of surgical pain after operation as assessed by visual analogue scale | 5 days after operation
  Visual analogue scale (VAS 1-10, a continuum scale in which 0 represents "no pain" and and 10 represents "worst pain.")
Rescue doses of analgesics administered after operation | 5 days after operation
  Total doses of parenteral administered opioids, NSAIDs, COX-2 inhibitors

SECONDARY OUTCOMES:
Incidence of chronic post-surgical pain | 3 months after operation
  Pain that newly develops after operation and lasts >2 months and other causes of pain are excluded
Satisfaction of living after surgery as assessed by the HRQoL SF-12 | 3 months after operation
  Quality of life will be assessed by the HRQoL SF -12 Questionnaire, which consists a physical component summary (PCS) and a mental component summary (MCS). The rating scales range from yes-no to likert scales, and the final score of PCS and MCS will be calculated by an algorithm (QualityMetric's SF-12v1®). Scores range from 0 to 100, in which lower scores mean lower health related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- E-Da Hospital, Yanchao, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: No